CLINICAL TRIAL: NCT06000267
Title: Incidence of Difficult Airway and Identification of Relevant Anthropometric Factors in Pediatric Patients Scheduled for Elective Surgery
Brief Title: Incidence and Contributing Anthropometric Factors of Difficult Airway in Pediatric Surgical Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Childrens Hospital Belgrade (Other)
Responsible Party: Principal Investigator, Ivana Petrov Bojicic, Associate Professor, University Childrens Hospital Belgrade
Other Study IDs: UCHBelgrade
Record Dates: First submitted 2023-08-12; First posted 2023-08-21 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-09

CONDITIONS: Difficult Airway
Keywords: children; intubation; face mask ventilation; best oropharyngeal view
MeSH Terms: interventions — Intubation

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Intubation — All the patients will be ventilated with face mask and intubated before elective surgery

SUMMARY:
The goal of this prospective, observational study is to identify predictors of difficult mask ventilation, direct laryngoscopy and intubation in pediatric patients scheduled for elective surgery and to determine their incidence. As a final goal, the investigators will try to define new scoring system for difficult airway prediction. Participants will be pediatric patients age infant till school age. Participants will have their airway assessed one day before surgery by taking anthropometric measurements of face and neck. After iv anesthesia induction and application of muscle relaxant, the investigators will assess difficulty of face mask ventilation by using grading from 0-4. Direct laryngoscopy will be performed with Macintosh blade and experienced anesthesiologist will determine Cormack - Lehane score as well as intubation difficulty score (IDS).

DETAILED DESCRIPTION:
Participants will be divided into groups: up to 1 yrs of age, 1-2.9 yrs, 3-4.9, 5-6.9, and 7 yrs and older.

The investigators will test predictive value, sensitivity and specificity of anthropometric parameters used for airway assessment in pediatric patients, as well as gender, age, BMI, ASA score.

Anatomical parameters that will be measured the day before surgery: chin, inter - incisor gap, hyomental distance (HMD), hyoid - thyroid distance (HT), neck circumference, neck length, neck extension, lower lip to chin distance (LCD), tragus to chin distance (TMA), thyromental distance (TMD), sternomental distance (SMD).

Mallampati test will be performed in children older than 5 years and best oropharyngeal view (BOV) will be determined for younger children. Colorado Pediatric Airway Score (COPUR) will be calculated.

All patients will be premedicated with midazolam 0.5 mg/kg orally, 30 minutes before intervention or 0.1 mg/kg iv. Anesthesia induction will be intravenous: thiopentone 5 mg/kg or propofol 2.5 mg/kg, fentanyl 3 mcg/kg and non depolarizing muscle relaxant rocuronium 1 mg/kg or cis-atracurium 0.15 mg/kg. Face mask ventilation will be quantified as grade 0-4. Anesthesia maintenance will be intravenous or inhalatory depending on anesthesiologists decision. Patients will be intubated with Macintosh blade in the supine position, without additional elevation of occipital part of the head. Difficult laryngoscopy is defined as CL grade III and IV and they predict difficult endotracheal intubation. Intubation difficulty score will be used to asses intubation. Intubation difficulty will be defined by IDS - intubation difficulty score > 5.

Standard procedures will be performed in case of difficult mask ventilation and intubation.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric patients from one month to 14 years old scheduled for elective surgery in general endotracheal anesthesia.

Exclusion Criteria:

* Congenital syndromes which include difficult airway (Pierre Robin, Goldenhar syndrome, Treacher Collins syn, Down syn, Edwards, Arthrogryposis, Apart syn etc.), craniofacial dysmorphia, ENT, maxillofacial and cardiac surgery patients, patients with resent respiratory infections

Ages: 28 Days to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Patient will be divided in 5 groups according to age: infants, children from 1 - 2,9 years, 3 - 4,9 years, 5 - 6,9 years and older than 7 years.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2022-01-10 (Actual); Primary Completion 2023-10 (Estimated); Study Completion 2023-10 (Estimated)

PRIMARY OUTCOMES:
incidence of difficult mask ventilation and intubation | one year
  Determination of grade 3 and 4 of mask ventilation incidence in different age groups of children and incidence of difficult intubation defined as intubation difficultly score >5

SECONDARY OUTCOMES:
Identification of anthropometric parameters of face and neck which determine difficult airway in children | one year
  Identification of preoperative measurements of face and neck determining difficult face mask ventilation and intubation

CONTACTS AND LOCATIONS:
Overall Officials: Ivana Petrov, MD, Principal Investigator — University children hospital
Locations (1):
- University Children hospital, Belgrade, Serbia

IPD SHARING:
Plan to Share IPD: No